CLINICAL TRIAL: NCT00973232
Title: A Single-Centre, Open-Label, Randomised Study to Compare the Single Dose (Including the Effect of Food) and Multiple Dose Pharmacokinetic Profiles of Acetram Contramid® BID Tablets vs the Immediate-Release Tablet Reference Products Zaldiar® and Ultracet®
Brief Title: A Comparative Bioavailability/Food Effect Study of Immediate-Release and Extended-Release Tramadol HCl/Acetaminophen Combination Products Following Single-Dose and Multiple-Dose Administration in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 06CCL102
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Tramadol; Acetaminophen; combination; pharmacokinetics; bioavailability; Zaldiar; Ultracet; fed; fasted; single-dose; multiple-dose; healthy; volunteers; Healthy volunteers
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Acetaminophen; Tramadol; Ultracet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part A, Arm A (Experimental)
  Interventions: Drug: DDS-06C (650 mg acetaminophen and 75 mg tramadol HCl)
- Part A, Arm B (Experimental)
  Interventions: Drug: DDS-06C (650 mg acetaminophen and 75 mg tramadol)
- Part A, Arm C (Active Comparator)
  Interventions: Drug: Zaldiar®
- Part A, Arm D (Active Comparator)
  Interventions: Drug: Ultracet®
- Part B, Arm E (Experimental)
  Interventions: Drug: Two tablets of DDS-06C (650 mg acetaminophen and 75 mg tramadol HCl), multiple doses, under both fed and fasting conditions
- Part B, Arm F (Active Comparator)
  Interventions: Drug: Zaldiar®, multiple doses,(fed & fasting):
- Part B, Arm G (Active Comparator)
  Interventions: Drug: Ultracet®, multiple doses, (fed & fasting)

INTERVENTIONS:
Drug: DDS-06C (650 mg acetaminophen and 75 mg tramadol HCl) — DDS-06C (650 mg acetaminophen and 75 mg tramadol HCl: two tablets, single dose, total administered of 1300 mg acetaminophen/150 mg tramadol HCl under fasting conditions
  Arms: Part A, Arm A
Drug: DDS-06C (650 mg acetaminophen and 75 mg tramadol) — DDS-06C (650 mg acetaminophen and 75 mg tramadol HCl: two tablets, single dose, total administered of 1300 mg acetaminophen/150 mg tramadol HCl under fed conditions
  Arms: Part A, Arm B
Drug: Zaldiar® — Zaldiar® (325 mg acetaminophen and 37.5 mg tramadol HCl): two tablets; dose of 650 mg acetaminophen/75 mg tramadol HCl administered at Time = 0 hr (fasting)and second dose at Time = 6 hr (fed) Ultracet® (325 mg acetaminophen and 37.5 mg tramadol HCl)
  Arms: Part A, Arm C
Drug: Ultracet® — Ultracet® (325 mg acetaminophen and 37.5 mg tramadol HCl)two tablets; dose of 650 mg acetaminophen/75 mg tramadol HCl administered at Time = 0 hr (fasting)and second dose at Time = 6 hr (fed) Ultracet® (325 mg acetaminophen and 37.5 mg tramadol HCl)
  Arms: Part A, Arm D
Drug: Two tablets of DDS-06C (650 mg acetaminophen and 75 mg tramadol HCl), multiple doses, under both fed and fasting conditions — Two tablets of DDS-06C, twice daily at 12-hour intervals under fed conditions for the first 4 days, then under fasting conditions for the 5th day. The total daily dose administered was 2600 mg Acetaminophen/300 mg tramadol HCl
  Arms: Part B, Arm E
Drug: Zaldiar®, multiple doses,(fed & fasting): — Two tablets of Zaldiar®, 4 times daily at 6-hour intervals under fed conditions for the first 4 days, then under fasting conditions for the 5th day. The total daily dose administered was 2600 mg Acetaminophen/300 mg tramadol HCl
  Arms: Part B, Arm F
Drug: Ultracet®, multiple doses, (fed & fasting) — Two tablets of Ultracet®, 4 times daily at 6-hour intervals under fed conditions for the first 4 days, then under fasting conditions for the 5th day. The total daily dose administered was 2600 mg Acetaminophen/300 mg tramadol HCl
  Arms: Part B, Arm G

SUMMARY:
The objectives of this two-part study were to compare the single-dose and multiple-dose pharmacokinetics of extended release and immediate-release fixed combination formulations containing tramadol-HCl/acetaminophen and to evaluate the effect of food on the extended-release formulation.

DETAILED DESCRIPTION:
* To compare the single (Part A) and multiple dose (Part B) pharmacokinetic profiles and bioavailability of DDS-06C tablets with the immediate-release tablet reference products Zaldiar® and Ultracet®.
* To assess the effect of food on the pharmacokinetic profile of DDS-06C tablets following administration of a single oral dose.
* To monitor and record all adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 18-55 years inclusive with body mass index (BMI) between 18-30 kg/m2
* Healthy as determined by pre-study medical history, physical examination and 12-lead ECG
* Clinical laboratory tests within the reference ranges or clinically acceptable to the Investigator
* Negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening
* Negative for drugs of abuse and alcohol at screening and admission
* Non-smokers for at least 3 months preceding screening
* If female, were not currently pregnant or breast feeding and were using medically acceptable methods of contraception and if male, were themselves and their female partners using medically acceptable methods of contraception
* Able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria
* Female subjects who were pregnant, trying to become pregnant, lactating or not using acceptable methods of contraception
* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders
* Clinically relevant surgical history
* Clinically relevant family history
* History of relevant atopy
* History of relevant drug hypersensitivity
* History of alcoholism
* History of drug abuse
* Male subjects who consumed more than 21 units of alcohol a week and female subjects who consumed more than 14 units of alcohol a week
* Significant infection or known inflammatory process on screening
* Acute gastrointestinal symptoms at the time of screening and/or admission (e.g. nausea, vomiting, diarrhoea, heartburn)
* Acute infection such as influenza at the time of screening or admission
* Use of prescription drugs within 7 days of first dosing, unless agreed as non clinically relevant by the Principal Investigator and Sponsor
* Use of over-the-counter medication excluding routine vitamins but including mega dose vitamin therapy within 14 days of first dosing, unless agreed as non clinically relevant by the Principal Investigator and Sponsor
* Use of any investigational drug or participation in any clinical trial within 3 months of their first dosing
* Donation or receipt of any blood or blood products within the previous 3 months prior to first dosing
* Vegetarians, vegans or having medical or cultural dietary restrictions.
* Inability to communicate reliably with the Investigator.
* Subjects who were unlikely to co-operate with the requirements of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Rate and extent of exposure | 0 to 36 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, Principal Investigator — Guy's Drug Research Unit, Quintiles Ltd
Locations (1):
- Guy's Drug Research Unit, Quintiles Ltd, London, United Kingdom